CLINICAL TRIAL: NCT04772066
Title: Evaluation of Tools to Assess Medication Adherence
Brief Title: Tools to Assess Medication Adherence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0662
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Medication Adherence
Keywords: Medication Adherence; Clinical Pharmacist; Self-reported scale
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non adherent patients: Non adherent patients
  Interventions: Other: Measure of medication adherence
- Adherent patients: Adherent patients
  Interventions: Other: Measure of medication adherence

INTERVENTIONS:
Other: Measure of medication adherence — Measure of medication adherence

SUMMARY:
The issue of medication adherence (MA) has long been undestimated but is now growing interest due to both the increase of patients with chronic diseases and the aging of the population. According to the World Health Organization, only 50% of patients with chronic illnesses correctly follow physician's prescriptions in developed countries. Beyond the individual consequences that failure to adherence can engender (increased morbidity, mortality and hospitalizations), this concept also encompasses a collective dimension (risk of transmission of infectious diseases and increased health care costs). Today, improving MA would have more impact on human health than developping new medical therapies. That's why detecting non-adherence constitutes a major public health issue in which pharmacists play a significant role through medication reconciliation and patients' education.

The methods wildly used are based on indirect measurement: questionnaires completed by the patient himself or the Medication Possession Ratio (MPR). Each method has its own advantages and disadvantages, but none is considered as the gold standard. The Montpellier University Hospital set up a MA self-report scale ranging from 0 (low) to 10 (high adherence) in the various care units where the clinical pharmacy activity is deployed.

The purpose of this study was to assess the MA according to this numerical scale and the MPR calculation, and evaluate the correlation between these two methods.

ELIGIBILITY:
Inclusion criteria:

- Subjects aged over 18 years old, admitted in a care unit of Montpellier University Hospital where the clinical pharmacy activity is deployed

Exclusion criteria:

- Subjects without any medication therapy at home

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of patients admitted in Montpellier University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported MA according to self-reported medication adherence scale | 1 day
  Self-reported MA according to self-reported MA scale : The self-report scale ranges from 0 (low) to 10 (high adherence)
MA according to Medication Possession Ratio (MPR) calculation | 1 day
  MA according to Medication Possession Ratio (MPR) calculation

SECONDARY OUTCOMES:
Number of patients with medication non-adherence according to self-reported MA scale and MPR calculation | 1 day
  Number of patients with medication non-adherence according to self-reported MA scale and MPR calculation
Variables associated with medication non-adherence | 1 day
  Variables associated with medication non-adherence

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, PharmD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC